CLINICAL TRIAL: NCT05426161
Title: The Effect of Subcutaneous Injection of Botulinum Toxin A on Chronic Wound Pain in Lower Extremities, a Prospective Exploratory Study
Brief Title: The Effect of Subcutaneous Injection of Botulinum Toxin A on Chronic Wound Pain in Lower Extremities
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Lubna Sabah, MD, Prinicipal Investigator, MD, Bispebjerg Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Botox-01
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Chronic Pain; Lower Extremity Wound
Keywords: Botulinum toxin A
MeSH Terms: conditions — Chronic Pain | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: A single-center, prospective, exploratory study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Botulinum Toxin A (Experimental): Open-label study
  Interventions: Drug: Botulinum Toxin A

INTERVENTIONS:
Drug: Botulinum Toxin A — Botulinum Toxin A (10 units per cm2 wound areal) will be injected subcutaneously around the wound (1-2 cm from wound edge) maximum 200 units at each injection time.The total dose of BoNTA is maximum 400 units. Patient will receive one or two treatments in total.

SUMMARY:
The aim of the study is to investigate the effect of subcutaneous administration of Botulinum toxin A on wound pain, wound healing and safety of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Lower extremity ulcer ≥ 4 weeks.
3. Ulcer area ≥ 1,5 cm2 and ≤ 20 cm2
4. Patients with neuropathic pain related to the ulcer (daily VAS pain scores ≥ 30 mm at rest and DN4 score ≥ 4).
5. Normal monofilament and vibration test in lower extremities.
6. Patients who can fill out pain diary correctly.
7. Written informed consent to participate in the study after having fully understood the contents of the protocol and restrictions.

Exclusion Criteria:

1. Infection at injection site. 2. Hypersensitivity to botulinum toxin A. 3. Peripheral neuropathy. 3. Diabetic foot ulcer. 4. Unstable critic peripheral ischemia judged by investigator 5. Exposed capsule, tendon, muscle or bone in the ulcers. 6. Tunnelling, undermining or sinus tracts. 7. Disorders of the neuromuscular junction (e.g. Myasthenia). 8. Topical analgesic (e.g Biatain ibu or Lidocain) within 7 days before inclusion.

9. Pregnant or lactating woman and woman with childbearing potential but does not use contraception.

10. Judgment by the investigator that the patient is not suited for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Proportion of patients reaching a reduction in mean visual analog scale (VAS) > 20 mm (at rest) in dynamic pain scores at study day 21 or 41 | 3 to 6 weeks after first injection of Botulinum toxin a
  At study day 0 the mean VAS will be calculated at rest for D-2-0 and at D21 or D41 mean VAS will be calculated for D19-21 or D39-41

SECONDARY OUTCOMES:
Absolute and percentage change in the area of hyperalgesia and allodynia | 3 to15 weeks after first injection of Botulinum toxin a.
  Area of hyperalgesia and allodynia will be assessed at D0, D21/41 and D90/110
Absolute and percentage change of the ulcer area. | Throughout the trial (12-15 weeks)
  The ulcer size will be measured at every visit with study day 0 as baseline.
Clinical improvement of the wound healing process | Throughout the trial (12-15 weeks)
  Semi-quantitatively measured (major improvement, minor improvement, status quo or worsening)
Therapeutic doses of Botulinum toxin a to treat wound pain | 3 and 6 weeks after first injection
  Number of patients who need a second injection of Botulinum toxin a on study D21 if mean VAS (D19-21) are similar (± 10 %) to the pre-injection mean VAS at D0
Incidence of Treatment-Emergent Adverse Events | Throughout the trial (12-15 weeks)
  All clinical adverse events will be assessed and recorded.
Exploratory measurement: Changes in the levels of cytokines and pain related substances in the wound fluid before and after injection with Botulinum toxin a | Analysis within 1 year after study completion
  Changes in the levels of cytokine and pain related substances will be quantified over time (throughout the trial). Prospects to analyse i.g ( IL-6, NGF, IL-1β) with either MSD,Luminex or ELISA.
  The results will be expressed as pg/ mg.

OTHER OUTCOMES:
Wound status- Degree of inflammation, granulation tissue, necrosis/slough, exudation and infection. | Throughout the trial (12-15 weeks)
  Semi-quantitatively measured (Absent/Low < 25 %, Mild 25-50 %, Moderate 51-75 %, High > 75%)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Francis Thomsen, Professor, Study Director — Department of Dermatology and Copenhagen Wound Healing Center, Bispebjerg Hospital
Locations (1):
- Department of Dermatology and Copenhagen Wound Healing Center, Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No